CLINICAL TRIAL: NCT07246512
Title: Comparison Between MTA and TotalFill® BC-RRM Fast Set Putty for Retrograde Filling in Apical Surgery: Randomized Non-inferiority Clinical Trial.
Brief Title: A Comparative Analysis of Biomaterials for Retrograde Filling in Apical Surgery.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Peñarrocha Oltra, Full Professor, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1. UV-INV_ETICA-1427893
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Periapical Lesion
Keywords: periapical lesion; endodontic failure; apical surgery; retrograde filling; periapical healing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MTA (Mineral Trioxide Aggregate) (Active Comparator): Patients undergoing apical surgery treated with retrograde obturation using Mineral Trioxide Aggregate (MTA).
  Interventions: Device: Mineral Trioxide Aggregate
- BioCeramic Root Repair Material Fast Set Putty (BCRRM) (Experimental): Patients undergoing apical surgery treated with retrograde obturation using BioCeramic Root Repair Material Fast Set Putty (BCRRM).
  Interventions: Device: BioCeramic Root Repair Material Fast Set Putty.

INTERVENTIONS:
Device: Mineral Trioxide Aggregate — Trioxide Mineral Aggregate as a retrograde filling material has 3 basic properties: biocompatibility, impermeable sealing of the root canal and properties that facilitate its clinical use. It has excellent properties that contribute to the healing of the periapical lesion.
  Other Names: MTA; ProRoot® MTA
  Arms: MTA (Mineral Trioxide Aggregate)
Device: BioCeramic Root Repair Material Fast Set Putty. — BioCeramic Root Repair Material (BCRRM) is a pre-mixed, easy to handle material that has demonstrated properties equivalent to MTA in terms of periapical lesion healing.
  Other Names: BCRRM; TotalFill® BC-RRM Fast Set Putty
  Arms: BioCeramic Root Repair Material Fast Set Putty (BCRRM)

SUMMARY:
The aim of this study is to compare two biomaterials used for retrograde obturation during apical surgery. This surgery is indicated in healthy patients when root canal treatment (endodontics) has failed to eliminate a periapical lesion (a persistent infection in the root of the tooth).

The main question it seeks to answer is:

- Is TotalFill® BC-RRM Fast Set Putty more effective than ProRoot® MTA in periapical surgery in terms of the degree of healing?

The study will include patients who need this type of surgery and meet specific clinical criteria. Each patient will have one of the two materials applied as part of the standard surgical procedure. Subsequently, clinical and radiographic follow-up will be performed to assess the degree of healing of the periapical lesion with a 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients giving consent for surgical intervention, for radiographic evaluation with HCT preoperatively and at least one more time after 12 months, and for participation in the study.
* Medical history not relevant to the diagnosis and surgical treatment (ASA classes I and II).
* Previous non-surgical endodontic treatment or retreatment with clinical and/or radiographic evidence of persistence or recurrence of apical periodontitis. The minimum time since the last non-surgical treatment shall be 6 months.
* Teeth not previously treated with periapical surgery.
* Lesion less than 10 mm in diameter.
* Restorable teeth.
* Periodontally sound teeth or teeth with treated periodontal pathology (mobility 1, probing depth < 5mm).
* Teeth with no root resorption.

Exclusion Criteria:

* Teeth with vertical fracture.
* Teeth with root perforation.
* Lesions associated with an apicomarginal defect.
* Tunnel lesions.
* Technical errors during surgery that may compromise the outcome.
* Lack of integrity of the dentine walls surrounding the retrograde filling detected with the endoscope.
* Wound dehiscence.
* Postoperative infection.
* Follow-up less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Periapical lesion healing assessed by CBCT using 3D PENN criteria. | 12 months post-surgery
  Periapical healing will be evaluated using cone-beam computed tomography (CBCT) at 12 months after periapical surgery. Lesion volume or dimensions will be measured and the percentage of reduction will be calculated. Based on these measurements, healing will be classified according to the 3D PENN CBCT criteria into complete, limited, uncertain, or unsatisfactory healing. A comparison will be made between ProRoot® MTA versus TotalFill® BC-RRM Fast Set Putty as retrograde filling materials.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Considerations about sharing individual participant data are ongoing. Any future data sharing will adhere to all institutional policies to ensure participant confidentiality.